CLINICAL TRIAL: NCT05706636
Title: T Central Memory Cells in Early Localized Non-Segmental Vitiligo and the Effect of Treatment
Brief Title: T Central Memory Cells in Early Localized Non-Segmental Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mogawer, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V-1-23
Record Dates: First submitted 2023-01-21; First posted 2023-01-31 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Vitiligo
Keywords: early localized vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Floderm topical cream

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early localized vitiligo on topical treatment (Active Comparator): Cases will only receive topical steroids/ calcineurin inhibitors and targeted phototherapy
  Interventions: Drug: Topical cream; Device: targeted phototherapy
- Early localized vitiligo on topical and systemic treatment (Active Comparator): Cases will receive oral mini-pulse steroids, topical steroids/ calcineurin inhibitors and targeted phototherapy
  Interventions: Drug: oral mini pulse; Drug: Topical cream; Device: targeted phototherapy

INTERVENTIONS:
Drug: oral mini pulse — 5mg / week oral dexamethasone
  Arms: Early localized vitiligo on topical and systemic treatment
Drug: Topical cream — topical fluticasone cream for body lesions and topical tacrolimus for face lesions
Device: targeted phototherapy — twice weekly targeted excimer light sessions

SUMMARY:
Assessing the level of circulating TCMs (cluster of differentiation (CD) 8+, CD3+,C- chemokine receptor (CCR)7, cluster of differentiation 45 receptor (CD45R) cells) in early localized vitiligo cases prior to treatment and after treatment in comparison to healthy controls. This, in turn, would provide insights regarding the role of TCMs in vitiligo and the role of early treatment in halting disease progression and autoimmune memory formation that accounts for high recurrence rate of vitiligo

DETAILED DESCRIPTION:
Assessing the level of circulating TCMs (CD8+ CD3+ CCR7+ CD45RO+ cells) in early localized vitiligo cases where samples will be processed and stained for CD8, CD3, CCR7, . CCR7, CD45R. Multi-parametric flow cytometry will be used to quantify CD3+ve, CD8+ve, CCR7+ve, CD45RO+ve TCM cells percentage, which will be expressed as a percentage from the total lymphocyte gate. This will be done prior to treatment and after treatment and will be compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with vitiligo localized to one anatomical area, of ≤ 6 months' duration

Exclusion Criteria:

* Patients who received treatment of any type (topical or systemic) within the last 3 months

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
comparing level of circulating central memory T cells (TCM) in early localized vitiligo cases to healthy controls | 6 months
  comparing TCM levels in early localized vitiligo cases prior to and after treatment to healthy controls
percent change in the level of circulating central memory T cells (TCM) in early localized vitiligo cases after treatment | 6 months
  assessing the level of circulating central memory T cells (TCM) in early localized vitiligo cases after treatment and calculating percent change in their levels
comparing percent change in the level of circulating central memory T cells (TCM) in early localized vitiligo cases after treatment in those receiving systemic treatment to those receiving only topical treatment | 6 months
  assessing the level of circulating central memory T cells (TCM) in early localized vitiligo cases after treatment and calculating percent change in their levels in those receiving systemic treatment to those receiving only topical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Samia Esmat, MD, Study Chair — Cairo University
Locations (1):
- Cairo university hospitals, dermatology outpatient clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participants' data that underlie reported results will be shared upon request, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 12 months after article publication
Access Criteria: Controlled Access:
  Researchers who provide a methodologically sound proposal will be allowed to access data to achieve aims in the approved proposal